CLINICAL TRIAL: NCT07299084
Title: A Study to Evaluate the Effect of Fasting Duration and Temporary Withholding of Tirzepatide on Retained Gastric Contents Using Gastric Ultrasound in Participants With Type 2 Diabetes Mellitus and Participants With Overweight or Obesity Without Type 2 Diabetes Mellitus
Brief Title: A Study to Evaluate the Effect of Fasting Duration and Tirzepatide Withholding on the Amount of Food and Fluid in the Stomach in Participants With Type 2 Diabetes Mellitus and Participants With Overweight or Obesity Without Type 2 Diabetes Mellitus
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 27358; I8F-MC-GPJE (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-12-10; First posted 2025-12-23 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Diabetes Mellitus, Type 2; Overweight; Obesity
Keywords: Point of Care Ultrasound (POCUS)
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Overweight; Obesity | interventions — Tirzepatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Participants with Type 2 Diabetes (Experimental): Participants will receive tirzepatide subcutaneously (SC)
  Interventions: Drug: Tirzepatide
- Participants with Overweight or Obesity Without Type 2 Diabetes (Experimental): Participants will receive tirzepatide SC
  Interventions: Drug: Tirzepatide

INTERVENTIONS:
Drug: Tirzepatide — Administered SC
  Other Names: LY3298176

SUMMARY:
The purpose of this study is to evaluate how fasting and stopping the use of tirzepatide affects the amount of food and drink that stays in the stomach after a meal. Ultrasound will be used to check the stomach content after a test meal.

ELIGIBILITY:
Inclusion Criteria:

* Meet one of the following criteria:

  * Have type 2 diabetes
  * Have obesity
  * Have overweight with at least one health issue related to weight but without type 2 diabetes

Exclusion Criteria:

* Have a condition that affects how their stomach empties
* Have had weight loss surgery
* Have type 1 diabetes
* Have any major medical conditions or histories that could interfere with the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Lack of Gastric Content Retention Post-Solid Test Meal | Baseline, Day 171 (at 6, 8, 12, 18 and 24 hours after baseline or Day 170 solid test meal)

SECONDARY OUTCOMES:
Percentage of Participants with Lack of Gastric Content Retention Post-Liquid Test Meal | Day 178 (at 6, 8, 12, 18 and 24 hours after Day 177 liquid test meal)
Amount of Gastric Content Volume Post-Liquid Test Meal | Day 178 (at 6, 8, 12, 18 and 24 hours after Day 177 liquid test meal)
Amount of Gastric Content Volume Post-Solid Test Meal | Baseline, Day 171 (at 6, 8, 12, 18 and 24 hours after baseline or Day 170 solid test meal)
Percentage of Participants with Lack of Gastric Content Retention Post-Solid Test Meal After Discontinuation of Tirzepatide | Baseline through 8 days after discontinuation of tirzepatide at 6, 8, 12,18 and 24 hours
Percentage of Participants with Grades 0, 1, and 2 from Antrum Grading Scale Post-Solid Test Meal | Baseline, Day 171 (at 6, 8, 12, 18 and 24 hours after baseline or Day 170 solid test meal)
Percentage of Participants with Grades 0, 1, and 2 from Antrum Grading Scale Post-Liquid Test Meal | Day 178 (at 6, 8, 12, 18 and 24 hours after Day 177 liquid test meal)]
Percentage of Participants with Grades 0, 1, and 2 from Antrum Grading Scale After Discontinuation of Tirzepatide | Baseline through 8 days after discontinuation of tirzepatide at 6, 8, 12,18 and 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Lilly Centre for Clinical Pharmacology, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Study to Evaluate the Effect of Fasting Duration and Tirzepatide Withholding on the Amount of Food and Fluid in the Stomach in Participants With Type 2 Diabetes Mellitus and Participants With Overweight or Obesity Without Type 2 Diabetes Mellitus — https://trials.lilly.com/en-US/trial/677436